CLINICAL TRIAL: NCT01453699
Title: Bereavement in Children, Adolescents and Young Adults. - A Study of Health and Psychosocial Well-being in Adults Who Have Experienced Early Parental Death
Brief Title: Long-term Consequences of Bereavement in Children, Adolescents and Young Adults
Status: Completed | Type: Observational
Sponsor: Danish Cancer Society (Other)
Collaborators: Statens Serum Institut (Other); Center for Crisis Psychology (Unknown); Counselling and Research Center for Grieving Children, Teens and Young Adults (Unknown); Children´s Welfare (Unknown)
Responsible Party: Principal Investigator, Christoffer Johansen, Head of Department of Psychosocial Cancer Research, Danish Cancer Society
Other Study IDs: 1-2009; 7134-08 (Other Grant/Funding Number: TrygFonden); 2009-41-3506 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2011-10-11; First posted 2011-10-18 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Bereavement
Keywords: Bereavement; early parental death; grief; affective disorders; depression, depressive symptoms; socioeconomic factors; suicide; attempted suicide; antidepressive agents; cardiovascular diseases; quality of life; Long-term health effects; Socioeconomic outcomes; Psychosocial well-being
MeSH Terms: conditions — Parental Death; Mood Disorders; Depression; Suicide; Suicide, Attempted; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine how the death of a parent as a child, adolescent or young adult affects health and psychosocial wellbeing in adult life and to evaluate the impact in adult life of counseling to children, adolescents and young adults who lost a parent.

DETAILED DESCRIPTION:
Early parental death experienced by 4% of the children in Western countries, is considered to be the most stressful and potentially harmful childhood life event and the health consequences may depend on the nature of the bereavement (e.g. relationship with bereaved), as well as by interpersonal (e.g. social support), intrapersonal (e.g. age and genetics), appraisal and coping factors. Studies have shown that children and adolescents have a greater risk of getting a psychiatric diagnose as well as psychological and social problems. Despite of the obvious consequences of losing a parent, there is a lack of systematic studies on the consequences later in life as well as studies that evaluate the counseling possibilities the children and adolescents are offered.

The study will investigate:

1. Long-term health effects of experiencing parental death as a child adolescent or young adult. Focus will be on psychiatric outcomes including depression, severe cardiovascular disease, suicide, suicide attempts, psychological well-being and health related behavior.
2. Long term effects of experiencing parental death as a child, adolescent or young adult on socioeconomic outcomes as education, employment, marital status/ cohabitation status and number of children/age when having children.
3. The long-term psychosocial and behavioral impact of psychological intervention programmes to children, adolescents and young adults who have experienced the death of a parent. Focus will be on: Depressive symptoms, quality of life, posttraumatic stress disorder, life style, relationship functioning, grief and spirituality.

A nationwide register based cohort of people born in Denmark will be established. Long-term health effects and socioeconomic outcomes of experiencing parental death will be based on nationwide clinical and administrative registries. Exposure is defined as experiencing the death of a parent before age 30. The long-term psychosocial and behavioral impact of psychological intervention programmes will be based on a combination of questionnaire data and data from registries.

The part of the study using data from registries will be based on the nationwide cohort. The questionnaire based part of the study will include 3 groups selected from the nationwide cohort:

1. Persons who have lost a parent and participated in intervention programmes (identified through counseling centers),
2. Persons who have lost a parent, and not participated in intervention programmes (randomly selected matched on age and gender) and
3. Persons who have not lost a parent (randomly selected matched on age and gender).

An invitation letter will be send to the 3 groups (5500 persons) by mail, and they will be asked to complete one questionnaire online.

ELIGIBILITY:
Inclusion Criteria:

* persons born in Denmark

Exclusion Criteria:

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nationwide population-based cohort (Denmark)
Sampling Method: Probability Sample
Enrollment: 1225660 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Hospitalization for affective disorder | Paticipants will be followed from age 15 until date of first hospitalization for an affective disorder, death, first emigration or end of follow up, an expected average of 12 years
  Danish Psychiatric Central Register
Use of antidepressive medication | Paticipants will be followed from age 20 until date of second independantly prescription of antidepressive medication, death, first emigration or end of follow up, an expected average of 9 years
  The Danish National Prescription Registry
Suicide | Paticipants will be followed from age 18 until date of suicide, other causes of death, first emigration or end of follow up, an expected average of 15 years
  Danish Register of Causes of Death
Severe cardiovascular disease | Paticipants will be followed from age 18 until date of first hospitalization for severe cardiovascular disease, death, first emigration or end of follow up, an expected average of 15 years
  The Danish National Patient Register
Education level | Participants will be followed from age 18 until highest attained educational level, death, first emigration or end of follow up, an average of 20 years
  The Register-based System of Demographics and Social Statistics in Denmark
Employment | Employment status at age 30, death, first emigration or end of follow-up, an expected average of 8 years.
  The Register-based System of Demographics and Social Statistics in Denmark
Quality of life | Participants will be answering the questionnaire once (not at a specifik age but between 18-40 years)
  SF-36, Self-reported questionnaire
Complicated grief | Participants will be answering the questionnaire once (not at a specifik age but between 18-40 years)
  Inventory of Complicated Grief/ Prolonged Grief Disorder (PG-13) and Centrality of Event Scale, Self-reported questionnaire
PTSD | Participants will be answering the questionnaire once (not at a specifik age but between 18-40 years)
  Harvard Trauma Questionnaire (HTQ), Self-reported questionnaire
Existentiality | Participants will be answering the questionnaire once (not at a specifik age but between 18-40 years)
  Posttraumatic Growth Inventory (PTGI, Self-reported questionnaire
Depressive symptoms | Participants will be answering the questionnaire once (not at a specifik age but between 18-40 years)
  The Center for Epidemiological Studies Depression Scale (CES-C)

SECONDARY OUTCOMES:
Relationship functioning | Participants will be answering the questionnaire once (not at a specifik age but between 18-40 years)
  Quality of relationship and intimacy, Self-reported questionnaire
Support when losing a parent | Participants will be answering the questionnaire once (not at a specifik age but between 18-40 years)
  Self-report items
Lifestyle (smoking, alcohol, exercise) | Participants will be answering the questionnaire once (not at a specifik age but between 18-40 years)
  Self-reported questionnaire
Coping | Participants will be answering the questionnaire once (not at a specifik age but between 18-40 years)
  Brief cope, Self-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Johansen, MD, PhD, DSc, Principal Investigator — Institute of Cancer Epidemiology, Danish Cancer Society; Charlotte W Appel, MSc, Study Chair — Institute of Cancer Epidemiology, Danish Cancer Society; Pernille E Bidstrup, PhD, Study Chair — Institute of Cancer Epidemiology, Danish Cancer Society; Henrik Hjalgrim, PhD, Study Chair — Statens Serum Institut
Locations (1):
- Department of Psychosocial Cancer Research, Institute of Cancer Epidemiology, Danish Cancer Society, Copenhagen, Denmark